CLINICAL TRIAL: NCT06164457
Title: Implementing Individualized Patient Reported Outcome Measures in Routine Care of Patients With Coronary Artery Disease: a Pilot Study
Brief Title: Implementing Individualized Patient Reported Outcome Measures in Routine Care of Patients With Coronary Artery Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Calgary (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: REB22-1370
Record Dates: First submitted 2023-12-01; First posted 2023-12-11 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-11

CONDITIONS: Coronary Artery Disease; Patient Acceptance of Health Care; Physician-Patient Relations
Keywords: coronary artery disease; patient reported outcome measures; cardiac science; communication assessment; quality improvement; feasibility
MeSH Terms: conditions — Coronary Artery Disease; Patient Acceptance of Health Care

STUDY DESIGN:
Intervention Model Description: Pre-post intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Patients in this group will attend their cardiology appointment as normal. No intervention present.
- Intervention Group (Experimental): Patients in this group will complete the ePROM patient survey in advance of their care visit.
  Interventions: Other: ePROM Survey

INTERVENTIONS:
Other: ePROM Survey — The APPROACH ePROM survey consists of several well validated PROM instruments, including the Seattle Angina Questionnaire 7-item version,[4] the EuroQol EQ5D-5L,[5] the Medical Outcomes Study Social Support Scale (8 item version),[6] the Patient Health Questionnaire 2-item and 9-item (PHQ2/9) depression screening tools[7], and the Self-Care of Coronary Heart Disease Inventory (SC-CHDI-V3).[8]
  Arms: Intervention Group

SUMMARY:
Investigators recently developed the APPROACH electronic patient reported outcome (ePROM) Survey and Clinician Report tools to collect individual results from online quality of life and health status surveys for patients with coronary heart disease, and report them back to their treating clinicians. This pilot interventional study uses a pre-post design to assess whether implementing the ePROM system into routine care is feasible and acceptable to patients and physicians, and to inform feasibility for a larger clinical trial. Specifically, the investigators aim to evaluate use of the ePROM Patient Survey and Clinician Report among eligible outpatients with known or suspected coronary artery disease and their cardiologists. Additionally, the investigators aim to determine if the use of the APPROACH ePROMs Clinician Report in routine medical encounters is acceptable (based on administrative burden, ease of use, and time required) to patients and clinicians, and supports effective communication for management of symptoms of coronary artery disease.

DETAILED DESCRIPTION:
Background

Electronic capture and reporting of patient reported outcome measures has the potential to improve patient-physician communication and the delivery of cardiac care for patients with chronic health conditions, including coronary artery disease.[1, 2] Input from both patients and clinicians was used to develop an ePROMs Patient Survey and a Clinician Report that summarizes and contextualizes the responses for patients with coronary artery disease. The investigators plan to perform a staged implementation of both aspects for patients attending cardiac catheterization labs in Alberta and evaluate the impact of this intervention on patient outcomes and use of health services in a randomized clinical trial. However, before proceeding with this large-scale trial, the investigators need to ensure that the intervention can be delivered effectively and assess its impact on the processes of care. This pilot study is designed to assess the perceived utility of the APPROACH ePROM Clinician Report in routine clinical care and to inform feasibility for a larger clinical trial.

Methods

Design: Prospective, pre-post intervention clinical study.

Setting: Outpatient cardiology practices in Alberta.

Study Design: In each cardiology practice, control group patients for 4 months or until 30 patients are enrolled, whichever is soonest. Once the control group enrolment target is reached in each practice, a formal training program covering the use of the ePROM Clinician Report will be delivered to each cardiologist. The practice will then transition to the intervention period. The intervention period will last 4 months or until 30 patients have been enrolled, whichever is soonest. Each patient will contribute a single visit, with no longitudinal follow-up.

Study Procedures - Control Period:

* Eligible patients in each participating clinician practice will be enrolled before providing the ePROMs intervention to establish the baseline level for several study measures, including satisfaction with care and level of communication (see Outcomes section below).
* Patient Screening and Recruitment. Patients who have an upcoming outpatient visit with a study cardiologist in the next 14-28 days will be screened by the cardiologist's office staff, who will obtain the patient's consent to be contacted by the research team. Research personnel will confirm study eligibility an\d then contact patients by telephone to explain the study and obtain their informed consent, as well as collecting baseline demographic (age, sex, ethnicity, education, employment), clinical (cardiac and non-cardiac medical history) and health literacy data. Patients will be asked to provide an email address for the purposes of receiving study communications.
* Pre-visit intervention: Control period patients will not receive the ePROMs survey to complete, and will not be further contacted by study personnel in advance of their cardiologist clinic visit.
* Post-visit data collection. Control period patients will be sent an electronic survey within 48 hours after their scheduled clinic visit, with a reminder phone call 4-7 days later to those who have not yet completed it. The survey will consist of the following components: Assessment of communication effectiveness for the visit, using the Communication Assessment Tool, and assessment of patient satisfaction with care at the study visit.

Study Procedures - Intervention period:

* Clinician Training. Participating cardiologists will provide informed consent for study participation and receive one-on-one training on the use and interpretation of the ePROMs Clinician Report prior to starting patient enrolment. Training will be conducted by research personnel and will include didactic components outlining the potential value of PROMs in routine care, interpretation of the report itself, and a list of potential resources for patients with non-cardiac concerns identified by the ePROMs tool. Research personnel will also provide information, training, and ongoing support to each participating cardiologist's office staff to ensure the success of screening and recruitment.
* Patient Screening and Recruitment. The initial screening, recruitment, and baseline data collection process will be identical to that for the control period.

Patient Survey. Consenting patients will be sent an email link to the APPROACH ePROM survey at least 7 days before their upcoming cardiologist appointment, and will be asked to complete it at least 72 hours before their appointment.

The APPROACH ePROM survey consists of several well validated PROM instruments, including the Seattle Angina Questionnaire 7-item version,[4] the EuroQol EQ5D-5L,[5] the Medical Outcomes Study Social Support Scale (8 item version),[6] the Patient Health Questionnaire 2-item and 9-item (PHQ2/9) depression screening tools[7], and the Self-Care of Coronary Heart Disease Inventory (SC-CHDI-V3).[8] To improve the survey completion rate, research staff will follow-up by telephone with the patient in the week before the clinic visit to offer support and a single system-generated reminder email will be sent 72 hours before the appointment. Patients who do not complete the survey in advance of the visit will be offered the opportunity to complete it while waiting for their appointment on a study-supplied iPad.

- Clinician Report. The research team will transmit the ePROM Clinician Report for each patient to the cardiologist's office in advance of the visit, using their preferred method (fax/email). Participating cardiologists will be sent weekly reminder emails to encourage them to use the reports, and to request any feedback on the study to date.

Sample size and statistical considerations This pilot study will use convenience sampling with no powered statistical inference testing planned. The investigators estimate that a total sample of 4 cardiologists and approximately 80 control group and 120 intervention group patients are needed to achieve the objectives of estimating the uptake and perceived acceptability / utility of both the ePROM Patient Survey and Clinician Report.

Expected outcomes

At the conclusion of this pilot study, the investigators will have an increased understanding of:

* A comparison of patient assessments of communication effectiveness and overall satisfaction of care before and after introduction of the ePROMs surveys and clinician reports.
* Both clinicians' and patients' perceptions about the acceptability and utility of ePROM Clinician Report as an adjunct to routine care for patients with coronary artery disease.
* The barriers and facilitators involved with implementing ePROMs Clinician Report in ambulatory care practices in Alberta.
* The overall and item-level completeness of the ePROM Patient Surveys.
* Preliminary estimates of the frequency with which the ePROM Clinician Report leads to a change in management of both cardiac and non-cardiac clinical concerns.

Limitations, Anticipated Risks and mitigation plan:

Recruitment of cardiology practices for the pilot. The research team includes cardiologists in both Calgary and Edmonton. The investigators will recruit from their colleagues, who have generally been supportive of other pilot activities in this area. The investigators will request basic information about their practice, including the frequency of clinics and case mix, prior to confirming their participation.

Recruitment of patients within clinics. The research team will provide significant training and ongoing support to the office staff at each clinic in order to encourage them to identify potential patients and perform the consent to contact activities.

Ensuring timely distribution of Clinician Report to clinics. The investigators will establish clinic-specific processes to ensure that the reports are received in the most convenient way for each participating clinic, with sufficient time for them to be incorporated into the medical record for review by the physician.

Reliance on self-report for measuring uptake of the clinician report. This study design does not have an objective measure of the use of the Clinician Report in each encounter. Directly observing encounters is not feasible. Therefore, the investigators are relying on patient self-report, which has limitations in terms of potential recall bias. The research team is mitigating this bias by performing the post-encounter survey as close to the visit as is feasible, and by comparing with a control period.

ELIGIBILITY:
Patient Inclusion Criteria:

* age at least 40 years.
* either (i) known coronary artery disease (defined as a history of myocardial infarction, percutaneous or surgical coronary revascularization, or documentation of obstructive coronary artery disease on previous invasive or CT angiography) or (ii) suspected coronary artery disease (defined as stable angina or anginal equivalent symptoms) as the reason for referral to a cardiologist.
* Able to communicate in English or be willing to have an English-speaking family member or friend assist with survey completion.
* Access to the internet, valid email address, and a web-enabled device, for survey completion.
* Upcoming outpatient visit with a study cardiologist in the next 14-28 day

Exclusion criteria:

- N/A, all inclusion criteria must be met to participate

Physician Inclusion Criteria: We will recruit 4 cardiologists to participate, 2 each from Alberta Health Services Edmonton and Calgary zones, including both academic and community practice settings. To be eligible, cardiologists will need to have an active outpatient practice including moderate to high volumes of patients being assessed and managed for coronary artery disease, and to be willing to commit to participating in all aspects of the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
ePROM usage metrics | Usage metrics will be collected during the intervention period (~4 months)
  data extract for the ePROM Patient Survey will be prepared, summarizing the proportion of patients who completed the survey, as well as scale-level and item-level missingness among completers. Quantitative data for each component subscale (SAQ-7, EQ5D-5L and VAS, MOS SSS, PHQ2/PHQ9, CAS) will be summarized. Our target is a ≥70% survey response rate, with ≥ 90% item-level completion rate among respondents.
Acceptability of the Clinician Report to clinicians | Post-visit surveys will be completed following every patient visit during the intervention period (~4 months), the exit interview will occur at the end of the intervention period.
  Participating cardiologists will be asked to complete an evaluation of their experience using the ePROM Clinician Report. This will be collected using a brief electronic survey administered after each study visit in the intervention period. This post-visit survey will be complemented by a single exit interview with participating physicians at study's end. The exit interview will assess the following using a semi-structured interview format with qualitative analysis.
Acceptability and utility of the ePROM Patient Survey and Clinician Report to patients | Patients will complete a post-visit survey following each visit during both the control and intervention period (~8 months).
  Participating patients will be sent an electronic survey within 48 hours after their scheduled clinic visit, with a reminder phone call 4-7 days later to those who have not yet completed it.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen B Wilton, MD, MSc, Principal Investigator — APPROACH Research Group, Libin Cardiovascular Institute, Cumming School of Medicine
Locations (2):
- Canada (2):
  - Cumming School of Medicine, University of Calgary, Calgary, Alberta
  - Department of Medicine, University of Alberta, Calgary, Alberta

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Greenhalgh J, Gooding K, Gibbons E, Dalkin S, Wright J, Valderas J, Black N. How do patient reported outcome measures (PROMs) support clinician-patient communication and patient care? A realist synthesis. J Patient Rep Outcomes. 2018 Sep 15;2:42. doi: 10.1186/s41687-018-0061-6. eCollection 2018 Dec. PMID 30294712
- [Background] Ishaque S, Karnon J, Chen G, Nair R, Salter AB. A systematic review of randomised controlled trials evaluating the use of patient-reported outcome measures (PROMs). Qual Life Res. 2019 Mar;28(3):567-592. doi: 10.1007/s11136-018-2016-z. Epub 2018 Oct 3. PMID 30284183
- [Background] Makoul G, Krupat E, Chang CH. Measuring patient views of physician communication skills: development and testing of the Communication Assessment Tool. Patient Educ Couns. 2007 Aug;67(3):333-42. doi: 10.1016/j.pec.2007.05.005. Epub 2007 Jun 18. PMID 17574367
- [Background] Chan PS, Jones PG, Arnold SA, Spertus JA. Development and validation of a short version of the Seattle angina questionnaire. Circ Cardiovasc Qual Outcomes. 2014 Sep;7(5):640-7. doi: 10.1161/CIRCOUTCOMES.114.000967. Epub 2014 Sep 2. PMID 25185249
- [Background] Feng YS, Kohlmann T, Janssen MF, Buchholz I. Psychometric properties of the EQ-5D-5L: a systematic review of the literature. Qual Life Res. 2021 Mar;30(3):647-673. doi: 10.1007/s11136-020-02688-y. Epub 2020 Dec 7. PMID 33284428
- [Background] Moser A, Stuck AE, Silliman RA, Ganz PA, Clough-Gorr KM. The eight-item modified Medical Outcomes Study Social Support Survey: psychometric evaluation showed excellent performance. J Clin Epidemiol. 2012 Oct;65(10):1107-16. doi: 10.1016/j.jclinepi.2012.04.007. Epub 2012 Jul 20. PMID 22818947
- [Background] Levis B, Sun Y, He C, Wu Y, Krishnan A, Bhandari PM, Neupane D, Imran M, Brehaut E, Negeri Z, Fischer FH, Benedetti A, Thombs BD; Depression Screening Data (DEPRESSD) PHQ Collaboration; Che L, Levis A, Riehm K, Saadat N, Azar M, Rice D, Boruff J, Kloda L, Cuijpers P, Gilbody S, Ioannidis J, McMillan D, Patten S, Shrier I, Ziegelstein R, Moore A, Akena D, Amtmann D, Arroll B, Ayalon L, Baradaran H, Beraldi A, Bernstein C, Bhana A, Bombardier C, Buji RI, Butterworth P, Carter G, Chagas M, Chan J, Chan LF, Chibanda D, Cholera R, Clover K, Conway A, Conwell Y, Daray F, de Man-van Ginkel J, Delgadillo J, Diez-Quevedo C, Fann J, Field S, Fisher J, Fung D, Garman E, Gelaye B, Gholizadeh L, Gibson L, Goodyear-Smith F, Green E, Greeno C, Hall B, Hampel P, Hantsoo L, Haroz E, Harter M, Hegerl U, Hides L, Hobfoll S, Honikman S, Hudson M, Hyphantis T, Inagaki M, Ismail K, Jeon HJ, Jette N, Khamseh M, Kiely K, Kohler S, Kohrt B, Kwan Y, Lamers F, Asuncion Lara M, Levin-Aspenson H, Lino V, Liu SI, Lotrakul M, Loureiro S, Lowe B, Luitel N, Lund C, Marrie RA, Marsh L, Marx B, McGuire A, Mohd Sidik S, Munhoz T, Muramatsu K, Nakku J, Navarrete L, Osorio F, Patel V, Pence B, Persoons P, Petersen I, Picardi A, Pugh S, Quinn T, Rancans E, Rathod S, Reuter K, Roch S, Rooney A, Rowe H, Santos I, Schram M, Shaaban J, Shinn E, Sidebottom A, Simning A, Spangenberg L, Stafford L, Sung S, Suzuki K, Swartz R, Tan PLL, Taylor-Rowan M, Tran T, Turner A, van der Feltz-Cornelis C, van Heyningen T, van Weert H, Wagner L, Li Wang J, White J, Winkley K, Wynter K, Yamada M, Zhi Zeng Q, Zhang Y. Accuracy of the PHQ-2 Alone and in Combination With the PHQ-9 for Screening to Detect Major Depression: Systematic Review and Meta-analysis. JAMA. 2020 Jun 9;323(22):2290-2300. doi: 10.1001/jama.2020.6504. PMID 32515813
- [Background] Vaughan Dickson V, Lee CS, Yehle KS, Mola A, Faulkner KM, Riegel B. Psychometric Testing of the Self-Care of Coronary Heart Disease Inventory (SC-CHDI). Res Nurs Health. 2017 Feb;40(1):15-22. doi: 10.1002/nur.21755. Epub 2016 Sep 30. PMID 27686630
- [Background] Davis FD. Perceived Usefulness, Perceived Ease of Use, and User Acceptance of Information Technology. MIS Quarterly. 1989; 13: 319-340.
- [Derived] Dalton M, Kruger D, Sajobi TT, Southern D, Wilson T, Har BJ, Graham MM, Wilton SB, James MT. Individualized Electronic Patient-Reported Outcome Measures As a Communication Aid in Outpatient Cardiology Care: A Study Protocol. CJC Open. 2025 Feb 18;7(5):678-685. doi: 10.1016/j.cjco.2025.02.009. eCollection 2025 May. PMID 40433203